CLINICAL TRIAL: NCT03400111
Title: Assessment of Low-level Laser Therapy Versus Paracetamol-caffeine Efficacy in Controlling Pain During Fixed Orthodontic Treatment and Their Role in Enhancing Oral-health-related Quality of Life: A Randomized Controlled Trial
Brief Title: The Role of Paracetamol-caffeine and Laser Irradiation on Controlling Pain and Discomfort During Orthodontic Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UDDS-Ortho-03-2018
Record Dates: First submitted 2018-01-09; First posted 2018-01-17 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Pain and Discomfort; Orthodontic Appliance Complication
MeSH Terms: conditions — Pain | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients in the first group will undergo active irradiation with low-level laser therapy but they will consume placebo tablets. Patients in the second group will consume real Panadol-extra tablets but they will be subjected to a placebo red-beam as if they are irradiated with a laser beam. Patients in the third group will be subjected to both placebo procedures (i.e. placebo red-beam and not low-level laser therapy and placebo tablets).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-level laser therapy (Experimental): Patients upper and lower jaws will be irradiated with low-level laser therapy at specific points on the alveolus around the teeth from the vestibular and lingual sides. This group of patients will be followed up till the end of treatment.
  Interventions: Radiation: low-level laser therapy
- Panadol-extra (Experimental): Patients will be given Panadol-extra (565 mg: 500 mg paracetamol and 65 mg caffeine) at specific time points to control pain and discomfort during orthodontic treatment. This group of patients will be followed up till the end of treatment.
  Interventions: Drug: Panadol-extra
- Traditional Treatment (No Intervention): Patients will not undergo any actual irradiation therapy or take any active tablets during orthodontic treatment.

INTERVENTIONS:
Radiation: low-level laser therapy — low-level laser therapy will be used to relieve pain and discomfort during orthodontic treatment at specific time points.
  Arms: Low-level laser therapy
Drug: Panadol-extra — Tablets of 565-mg Panadol-extra will be used at specific time points to control pain and discomfort
  Arms: Panadol-extra

SUMMARY:
Patients with class I malocclusion who have mild to moderate crowding will be treated in this study. The efficacy of low level laser therapy and Panadol-extra® in relieving pain due to orthodontic treatment will be assessed. The effect of these two interventions on oral-health related quality of life during all stages of orthodontic treatment will be explored, i.e. at the following stages: (1) separation between teeth, (2) archwire changing, (3) bonding of brackets, (4) removal of the fixed appliances.

There are three groups :

1. a group of patient being irradiated with low-level laser therapy (LLLT) at specific time points to relieve pain and discomfort.
2. a group of patient in which pain control will be accomplished by prescribing Panadol Extra tablets in a regular manner.
3. a group of patients in which nothing will be given to them during the course of treatment.

DETAILED DESCRIPTION:
The assessment of oral-health-related quality of life during the different stages of orthodontic treatment is probably unique in the literature.

The study will cover the different stages of orthodontic treatment from A to Z. In other words, patients will be followed up till the end of treatment at which fixed appliances are removed. Pain control will be accomplished in one arm using LLLT and in another arm by prescribing Panadol Extra®. A third group will be left without any medication or laser irradiation to serve as a control group.

ELIGIBILITY:
Inclusion Criteria:

* Class I malocclusion with mild to moderate crowding (2-5 mm of tooth-size-arch-length-discrepancy)..
* Good oral hygiene and periodontal health
* No need for any preparation for fixed orthodontic appliance.
* No severe skeletal discrepancy (i.e. Class I skeletal relationship).

Exclusion Criteria:

* Previous orthodontic treatment
* Patients with psychological abnormalities.
* Patients with systematic diseases or being treated from chronic pain or headache.

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Change in Levels of Pain and Discomfort_Separation | (1) one hour following insertion of separators, (2) 24 hours, (3) 2 days, (4) seven days, (5) next meeting which is expected to be within 14 to 21 days.
  Patients will be given a rating numeric scale (RNS) to show their level of pain and discomfort after performing the first step in orthodontic installation of the appliance, i.e. the separation stage where separators are placed between the molar teeth on both sides of the jaw and in both jaws. Separators are placed for seven days before cementing the bands (that surround the molar teeth).
Change in Levels of Pain and Discomfort_FirstArch | (1) one hour following insertion of separators, (2) 24 hours, (3) 2 days, (4) seven days, (5) next meeting which is expected to be within 14 to 21 days.
  Patients will be given a rating numeric scale (RNS) to show their level of pain and discomfort after banding the molars and bonding the rest of the dental arches. Brackets are to be placed and the first archwire will be engaged. Assessment will be made at this stage which is called 'First Arch Placement'.
Change in Levels of Pain and Discomfort_SecondArch | (1) one hour following insertion of separators, (2) 24 hours, (3) 2 days, (4) seven days, (5) next meeting which is expected to be within 14 to 21 days.
  Patients will be given a rating numeric scale (RNS) to show their level of pain and discomfort after inserting the second arch in the sequence of arches of the orthodontic treatment. Assessment will be made at this stage which is called 'Second Arch Placement'.
Change in Levels of Pain and Discomfort_ThirdArch | (1) one hour following insertion of separators, (2) 24 hours, (3) 2 days, (4) seven days, (5) next meeting which is expected to be within 14 to 21 days.
  Patients will be given a rating numeric scale (RNS) to show their level of pain and discomfort after inserting the third arch in the sequence of arches of the orthodontic treatment. Assessment will be made at this stage which is called 'Third Arch Placement'.
Change in Levels of Pain and Discomfort_FouthArch | (1) one hour following insertion of separators, (2) 24 hours, (3) 2 days, (4) seven days, (5) next meeting which is expected to be within 14 to 21 days.
  Patients will be given a rating numeric scale (RNS) to show their level of pain and discomfort after inserting the fourth arch in the sequence of arches of the orthodontic treatment. Assessment will be made at this stage which is called 'Fourth Arch Placement'.
Change in Levels of Pain and Discomfort_LastArch | (1) one hour following insertion of separators, (2) 24 hours, (3) 2 days, (4) seven days, (5) next meeting which is expected to be within 14 to 21 days.
  Patients will be given a rating numeric scale (RNS) to show their level of pain and discomfort after inserting the fifth (i.e. the last) arch in the sequence of arches of the orthodontic treatment. Assessment will be made at this stage which is called 'Last Arch Placement'.
Change in Levels of Pain and Discomfort_Debonding | (1) one hour following insertion of separators, (2) 24 hours, (3) 2 days, (4) seven days, (5) next meeting which is expected to be within 14 to 21 days.
  Patients will be given a rating numeric scale (RNS) to show their level of pain and discomfort after appliance removal (i.e. taking off all the braces and bands). Assessment will be made at this stage which is called 'Appliance Removal'.

SECONDARY OUTCOMES:
Change in oral-health-related quality of life_Separation | (1) one week following separation, (2) at the following clinical visit which is usually expected to occur within 14 to 21 days.
  Patients will be given a questionnaire to be filled after performing the first step in orthodontic installation of the appliance, i.e. the separation stage where separators are placed between the molar teeth on both sides of the jaw and in both jaws. Separators are placed for seven days before cementing the bands (that surround the molar teeth). This questionnaire is called Oral-Health-Impact-Profile with 14 items (OHIP-14) which can be filled with three minutes.
Change in oral-health-related quality of life_FirstArch | (1) one week following archwire engagement, (2) at the following clinical visit which is usually expected to occur within 14 to 21 days.
  Patients will be given a questionnaire to be filled after banding the molars and bonding the rest of the dental arches. Brackets are to be placed and the first archwire will be engaged. Assessment will be made at this stage which is called 'First Arch Placement'. The questionnaire to be used is called Oral-Health-Impact-Profile with 14 items (OHIP-14) which can be filled with three minutes.
Change in oral-health-related quality of life_SecondArch | (1) one week following archwire engagement, (2) at the following clinical visit which is usually expected to occur within 14 to 21 days.
  Patients will be given a questionnaire to be filled after inserting the second arch in the sequence of arches of the orthodontic treatment. Assessment will be made at this stage which is called 'Second Arch Placement'.The questionnaire to be used is called Oral-Health-Impact-Profile with 14 items (OHIP-14) which can be filled with three minutes.
Change in oral-health-related quality of life_ThirdArch | (1) one week following archwire engagement, (2) at the following clinical visit which is usually expected to occur within 14 to 21 days.
  Patients will be given a questionnaire to be filled after inserting the third arch in the sequence of arches of the orthodontic treatment. Assessment will be made at this stage which is called 'Third Arch Placement'.The questionnaire to be used is called Oral-Health-Impact-Profile with 14 items (OHIP-14) which can be filled with three minutes.
Change in oral-health-related quality of life_FourthArch | (1) one week following archwire engagement, (2) at the following clinical visit which is usually expected to occur within 14 to 21 days.
  Patients will be given a questionnaire to be filled after inserting the fourth arch in the sequence of arches of the orthodontic treatment. Assessment will be made at this stage which is called 'Fourth Arch Placement'.The questionnaire to be used is called Oral-Health-Impact-Profile with 14 items (OHIP-14) which can be filled with three minutes.
Change in oral-health-related quality of life_LastArch | (1) one week following archwire engagement, (2) at the following clinical visit which is usually expected to occur within 14 to 21 days.
  Patients will be given a questionnaire to be filled after inserting the fifth (i.e. the last) arch in the sequence of arches of the orthodontic treatment. Assessment will be made at this stage which is called 'Last Arch Placement'.The questionnaire to be used is called Oral-Health-Impact-Profile with 14 items (OHIP-14) which can be filled with three minutes.
Change in oral-health-related quality of life_Debonding | (1) one week following appliance removal, (2) at the following clinical visit which is usually expected to occur within 14 to 21 days.
  Patients will be given a questionnaire to be filled after appliance removal (i.e. taking off all the braces and bands). Assessment will be made at this stage which is called 'Appliance Removal'.

OTHER OUTCOMES:
Psychological General Well-being | One week before performing the first step in Orthodontic Appliance Installation (i.e. one week before separation)
  Patients will be requested to fill in the Psychosocial General Well-being Index (PGWBI) before the commencement of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Amer M Owayda, DDS, Principal Investigator — MSc student in Orthodontics, University of Damascus Dental School, Damascus, Syria; Mohammad Y Hajeer, DDS MSc PhD, Study Chair — Associate Professor of Orthodontics, Department of Orthodontics, University of Damascus Dental School, Damascus, Syria; Rashad T Murad, DDS MSc PhD, Study Director — Associate Professor of Toxins and Pharmaceutics , Faculty of Pharmacology, University of Damascus, Damascus, Syria
Locations (1):
- Department of Orthodontics, University of Damascus Dental School, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Artes-Ribas M, Arnabat-Dominguez J, Puigdollers A. Analgesic effect of a low-level laser therapy (830 nm) in early orthodontic treatment. Lasers Med Sci. 2013 Jan;28(1):335-41. doi: 10.1007/s10103-012-1135-y. Epub 2012 Jul 21. PMID 22814893
- [Background] Choi SH, Kim JS, Cha JY, Hwang CJ. Effect of malocclusion severity on oral health-related quality of life and food intake ability in a Korean population. Am J Orthod Dentofacial Orthop. 2016 Mar;149(3):384-90. doi: 10.1016/j.ajodo.2015.08.019. PMID 26926026
- [Background] Dominguez A, Velasquez SA. Effect of low-level laser therapy on pain following activation of orthodontic final archwires: a randomized controlled clinical trial. Photomed Laser Surg. 2013 Jan;31(1):36-40. doi: 10.1089/pho.2012.3360. Epub 2012 Dec 16. PMID 23240876
- [Background] Farzanegan F, Zebarjad SM, Alizadeh S, Ahrari F. Pain reduction after initial archwire placement in orthodontic patients: a randomized clinical trial. Am J Orthod Dentofacial Orthop. 2012 Feb;141(2):169-73. doi: 10.1016/j.ajodo.2011.06.042. PMID 22284284
- [Background] Gupta M, Kandula S, Laxmikanth SM, Vyavahare SS, Reddy SB, Ramachandra CS. Controlling pain during orthodontic fixed appliance therapy with non-steroidal anti-inflammatory drugs (NSAID): a randomized, double-blinded, placebo-controlled study. J Orofac Orthop. 2014 Nov;75(6):471-6. doi: 10.1007/s00056-014-0243-7. Epub 2014 Oct 31. PMID 25355194
- [Background] Kim WT, Bayome M, Park JB, Park JH, Baek SH, Kook YA. Effect of frequent laser irradiation on orthodontic pain. A single-blind randomized clinical trial. Angle Orthod. 2013 Jul;83(4):611-6. doi: 10.2319/082012-665.1. Epub 2012 Dec 14. PMID 23241006
- [Background] Long H, Wang Y, Jian F, Liao LN, Yang X, Lai WL. Current advances in orthodontic pain. Int J Oral Sci. 2016 Jun 30;8(2):67-75. doi: 10.1038/ijos.2016.24. PMID 27341389
- [Derived] Owayda AM, Hajeer MY, Al-Sabbagh R, Burhan AS, Darwich K, Aljabban O, Latifeh Y. A randomized controlled trial on the effectiveness of low-level laser therapy versus paracetamol-caffeine for pain control during overall orthodontic treatment. Sci Rep. 2025 Aug 22;15(1):30839. doi: 10.1038/s41598-025-16658-2. PMID 40847180